CLINICAL TRIAL: NCT05645406
Title: Evaluating Quality Performance of Extemporaneously Compounded Estrogen Hormone Products
Brief Title: Estrogen Hormone Products
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Audra Stinchcomb, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00100540
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Menopause
MeSH Terms: interventions — Estradiol; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Divigel 0.1% (Active Comparator): Divigel 0.1% (1.25 g of gel/dose)
  Interventions: Drug: Divigel 0.1% Topical Gel
- Compounded estradiol product (Active Comparator): Compounded estradiol product (equivalent to Divigel/dose)
  Interventions: Drug: Compounded estradiol product

INTERVENTIONS:
Drug: Divigel 0.1% Topical Gel — estradiol topical products
  Other Names: estradiol gel
  Arms: Divigel 0.1%
Drug: Compounded estradiol product — estradiol topical products
  Other Names: estradiol topical product
  Arms: Compounded estradiol product

SUMMARY:
The purpose is to determine if the two estradiol products can deliver similar amounts of estradiol after single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, who are of any ethnic background, between the age of 45 to 65 years old
2. Provide written informed consent before initiation of any of the study procedures
3. Able to adhere to the study restrictions and study schedule
4. Volunteer has mid thighs of at least 42 cm (16.5 in) in circumference to accommodate the products to be tested at an area of 400 cm2 per thigh
5. Volunteer has legs that measure ≥46 cm (18.1 in) in length from the iliac crest to the top of the patella or large enough to accommodate the products to be tested at an area of 400 cm2 per thigh with the subject being comfortable with the template placement
6. Volunteer deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination, and medication history
7. Negative urine drug screening test (cannabinoids, amphetamines, barbiturates, benzodiazepine, cocaine, methadone, opiates, PCP)
8. Have normal screening laboratories for white blood cells (WBC), hemoglobin (Hgb), platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), creatinine, alanine transaminase (ALT), and aspartate aminotransferase (AST)
9. Have normal screening laboratories for urine protein and urine glucose
10. Naturally postmenopausal (absence of periods for ≥ 1 year or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy (menopause induced by removal of ovaries)
11. Agree not to participate in another clinical trial/study or to participate in an investigational drug study for at least one month after the last procedure day
12. Agrees not to donate blood to a blood bank throughout participation in the study and for at least three months after last procedure day
13. Have a normal ECG; must not have the following to be acceptable: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block. (sinus rhythm is between 55-100 beats per minute)
14. Have normal vital signs:

    * Temperature 35-37.9°C (95-100.3°F)
    * Systolic blood pressure 90-165 mmHg
    * Diastolic blood pressure 60-100 mmHg
    * Heart rate 55-100 beats per minute
    * Respiration rate 12-20 breaths per minute

Exclusion Criteria:

1. Smokers/tobacco users (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, snuff, gum, patches, or electronic cigarettes)
2. Participation in any ongoing clinical drug trial/study
3. Hereditary skin disorders or any skin inflammatory conditions as reported by the volunteer or evident to the MAI
4. History of significant dermatologic cancers (e.g., melanoma, squamous cell carcinoma) except basal cell carcinomas that were superficial and did not involve the investigative sites
5. History as either reported by the volunteer or evident to the investigator of infectious disease or skin infection or of chronic skin disease (e.g., psoriasis, atopic dermatitis)
6. Use of medications/alternative treatments/natural products for menopausal symptoms within the last 30 days or during the study.
7. Use of some chronic prescription medications during the period 0 to 30 days; or over-the-counter medications (e.g. antihistamines, topical corticosteroids, creams, gels, or ointments on your legs) and short term (<30 days) prescription medications during the period 0-3 days before a procedure day vitamin and herbal supplements not included). Certain types of medications may not exclude volunteers from this study, for example; thyroid medications, allergy medication that is not a steroid, non-steroidal anti-inflammatory drugs (e.g., ibuprofen or naproxen), and lipid/cholesterol lowering drugs.
8. Active positive Hepatitis B, C and/or HIV serologies
9. Positive urine drug screening test
10. Use of estrogen-containing implants, topical, or oral products
11. Donation or loss of greater than one pint of blood within 60 days of entry to the study
12. Any prior allergies to estradiol and its products or other ingredients in the applied gel or cream
13. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within one month before enrollment in this study or expects to receive an experimental agent during the study
14. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the volunteer at an unacceptable risk of injury or render the volunteer unable to meet the requirements of the protocol
15. History of diabetes
16. Breast cancer or history of breast cancer
17. Undiagnosed abnormal genital bleeding
18. Estrogen-dependent neoplasia (tumor)
19. Active arterial thromboembolic disease (example, stroke or heart attack), or a history of these conditions
20. Active DVT (blood clots in deep vein such as lower leg, thigh, pelvis or can occur in arm), PE (blood clot in blood vessel; often leg), or history of these conditions
21. Hepatic (liver) impairment or disease
22. A history of Protein C, protein S, or antithrombin deficiency, or other known thrombophilic disorders (tendency to form blood clots)
23. At application site, volunteer has an obvious difference in skin color between thighs, presence of a skin condition, excessive hair, sunburn, raised moles and scars, open sores, scar tissue, tattoo, or coloration that would interfere with placement of products, skin assessment, or reactions to estradiol
24. BMI ≥32 kg/m2

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
PK | -1 through 12 hours for four consecutive days
  serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Audra Stinchcomb, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- General Clinical Research Center (GCRC) at the University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be shared via a published manuscript.